CLINICAL TRIAL: NCT06597110
Title: The Effects of Autonomous Sensory Meridian Response (ASMR) on Sleep Quality Improvement in Adolescents
Acronym: ASMR on sleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Kai Zhao, associate pfofessor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUST-2023-108; KF202202 (Other Grant/Funding Number: huazhong university of science and technology)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Insomnia; Sleep Quality
Keywords: adolescent sleep; ASMR; sleep intervention; sleep quality scale
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The study involved sixty participants, divided evenly into four groups: three intervention groups (A, B, C) and one control group. For five consecutive days, the intervention groups engaged in pre-sleep ASMR listening sessions lasting 10, 20, and 30 minutes, respectively. Sleep quality was evaluated using mobile application tools and the subjective Sleep Quality Scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- control group (No Intervention): participants with no ASMR intervention
- intervention group A (Experimental): participants engaged in pre-sleep ASMR listening sessions lasting 10 mins
  Interventions: Behavioral: listened to ASMR
- intervention group B (Experimental): participants engaged in pre-sleep ASMR listening sessions lasting 20 mins
  Interventions: Behavioral: listened to ASMR
- intervention group C (Experimental): participants engaged in pre-sleep ASMR listening sessions lasting 30 mins
  Interventions: Behavioral: listened to ASMR

INTERVENTIONS:
Behavioral: listened to ASMR — ASMR refers to a physiological sensation triggered by specific auditory stimuli.ASMR, characterized by low-frequency human voice and ambient sounds, has garnered significant attention across social media platforms, short and long-form video platforms, and podcasts, owing to its unique pleasurable and stimulating effects. listen to ASMR for 10mins.
  Other Names: listern; ASMR
  Arms: intervention group A; intervention group B; intervention group C

SUMMARY:
Background: This study explored the therapeutic impact of ASMR on sleep problems in high school students.

Methods: The study involved sixty participants, divided evenly into four groups: three intervention groups (A, B, C) and one control group. For five consecutive days, the intervention groups engaged in pre-sleep ASMR listening sessions lasting 10, 20, and 30 minutes, respectively. Sleep quality was evaluated using mobile application tools and the subjective Sleep Quality Scale.

DETAILED DESCRIPTION:
Background: In recent years, there has been a notable surge in sleep-related challenges among adolescents. The emergence of Autonomous Sensory Meridian Response (ASMR) content across various social media platforms has sparked interest in its potential to address these issues. This study explored the therapeutic impact of ASMR on sleep problems in high school students.

Methods: The study involved sixty participants, divided evenly into four groups: three intervention groups (A, B, C) and one control group. For five consecutive days, the intervention groups engaged in pre-sleep ASMR listening sessions lasting 10, 20, and 30 minutes, respectively. Sleep quality was evaluated using mobile application tools and the subjective Sleep Quality Scale.

ELIGIBILITY:
Inclusion Criteria:

* Haven't heard an ASMR trigger tone before.

Exclusion Criteria:

* heard an ASMR trigger tone before.

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-08-06 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | 0ne month
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire designed to assess sleep quality and disturbances over a one-month period. It consists of 19 questions covering various aspects of sleep, such as sleep duration, latency, efficiency, and disturbances. The responses are used to calculate a global score, with higher scores indicating poorer sleep quality. It's commonly used in clinical and research settings to evaluate sleep-related issues and their impact on overall health.

SECONDARY OUTCOMES:
effective sleep time | 0ne month
  effective sleep time

CONTACTS AND LOCATIONS:
Overall Officials: Huiping Zhang, doctor, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR